CLINICAL TRIAL: NCT01391260
Title: A Phase II Trial of Radiation Therapy Combined With Iressa in Patients With Locally Advanced Non-small Cell Lung Cancer With Harboring Active EGFR Mutations
Brief Title: Radiotherapy Combined With Iressa for EGFR Mutation Positive Patients With Locally Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ZhuGuangYing (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Zhejiang Cancer Hospital (Other); Fudan University (Other); Renmin Hospital of Wuhan University (Other); 307 Hospital of PLA (Other); Beijing Clinical Service Center (Other)
Responsible Party: Zhu Guangying, Beijing Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-S10-09
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Locally Advanced NSCLC; EGFR Mutation Positive; Radiotherapy combined Gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy Combined With Gefitinib (Experimental)
  Interventions: Other: Gefitinib

INTERVENTIONS:
Other: Gefitinib — Radiation Therapy: 3D-CRT/IMRT 95%PTV 60-66Gy, 1.8-2.0Gy/f,5f/w; Gefitinib: 250 mg, Qd, p.o;
  Other Names: Iressa

SUMMARY:
The purpose of this study is to access the effect and safety of radiotherapy combined whth Iressa for patients with locally advanced non-small cell lung cancer with harboring active EGFR mutations.

DETAILED DESCRIPTION:
Worldwide more than half a million new cases of lung cancer are diagnosed annually. About 80% of these tumours are of non-small cell histological type. Surgery is the treatment of choice, but only about 20% of tumours are suitable for potentially curative resection. Concurrent chemoradiotherapy is the standard treatment for locally advanced NSCLC. When Iressa was used in the first-line treatment of advanced NSCLC with EGFR mutations positive, the 12-month rates of progression-free survival were 24.9%. Therefore, we speculate that the EGFR mutations in patients with locally advanced NSCLC, Gefitinib combined with radiotherapy may be better than chemoradiotherapy. We design the study to access the effect and safety of radiotherapy combined whth Iressa for patients with locally advanced non-small cell lung cancer with harboring active EGFR mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-squamous NSCLC; Stage ⅢA-ⅢB(not suitable for surgery) or stage Ⅳ(only single-site single transfer );
* Untreated patients, or who completed ≤ 2 cycles of first-line chemotherapy (chemotherapy regimen: paclitaxel, docetaxel + cisplatin) within the previous month;
* Patients with tumor EGFR mutation positive (exon 19 deletion mutation or exon 21 L858R substitution mutation);
* Patients must be informed of the investigational nature of the study and must sign an informed consent form;
* Presence of at least one measurable/evaluable according to RECIST criteria.
* ECOG performance Status 0-2 ;
* Patients must have a life expectancy > 12 weeks;
* Patients with laboratory values as follows:WBC>4.0 x 109/L; ANC≥1.5 x 109/L; PLT≥100 x 109/L; HGB≥10 g/dL; CR≤1.5 x ULN; TBIL<1.5 x ULN; AST and ALT≤1.5 x ULN; LDH≤1.5 x ULN; AKP≤5 x ULN;
* FEV 1≥1.0L and >50% Corresponding normal values;
* Patient candidate to standard platinum-based chemotherapy;
* Patients must be nonpregnant and non-lactating.Patients of childbearing potential must implement an effective method of contraception during the study. All female Patients, except those who are postmenopausal or surgically sterilized, must have a negative pre-study serum or urine pregnancy test.

Exclusion Criteria:

* Any evidence of clinically active interstitial lung disease;
* Diagnosis of any other malignancy during the last 5 years, except for in situ carcinoma of cervix uterine and squamous cell carcinoma of the skin；
* Pregnancy or lactating；
* Serious concomitant infection;
* MI within preceding 6 months or symptomatic heart disease, including unstable angina, congestive heart failure or uncontrolled arrhythmia;
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (eg, unstable or uncompensated respiratory, cardiac, hepatic, or renal disease);
* Patients who are not suitable to participate in the trial according to researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Response rate (RR) | 1 year

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
Overall survival (OS) | 2 years
Quality of life (MD-Anderson questionnaire) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Guangying, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (6):
- China (6):
  - 307 Hosptial of PLA, Beijing, Beijing Municipality
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality
  - Renmin Hospital of Wuhan University, Hubei General Hospital, Wuhan, Hubei
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing